CLINICAL TRIAL: NCT07354854
Title: Evaluation of the Safety and Effectiveness of the Tri-staple Technology inThoracic Surgery Clinical Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ezisurg Medical Co. Ltd. (Other)
Collaborators: Jinhua Municipal Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JH-Lite-T
Record Dates: First submitted 2025-12-29; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer (Diagnosis)
MeSH Terms: conditions — Lung Neoplasms; Disease | interventions — Thoracic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ezisurg stapler (Experimental)
  Interventions: Device: thoracic surgery

INTERVENTIONS:
Device: thoracic surgery — thoracic surgery using the easyEndo™ Lite Linear Cuting Stapler for Single Use and Loading Unites for Single Use for tissue cutting and suturing.

SUMMARY:
The goal of this post-market clinical study is to evaluate the safety and effectiveness of the tri-staple technology in thoracic surgery. The main question it aims to answer is to validate its efficacy, safety and operationalperformance for lung applications.

Participants will undergoing thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years old, male or female;
2. Subjects are scheduled to undergo open or thoracoscopic puimonary surgery with any surgicalprocedure;
3. The surgery is performed using the easyEndotm Lite Linear Cuting Stapler for Single Use andLoading Unites for Single Use for tissue cutting and suturing.

Exclusion Criteria:

1. Non-elective surgery;
2. Previous surgical operation on the ipsilateral lung;
3. Pregnant or lactating women;
4. Patients who, in the judgment of the investigator, are unsuitable to participate in the study for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Anastomosis success rate | Perioperative/Periprocedural
  Tissue transection andanastomosis are performed during the procedure, and the device is withdrawn after a successful trigger, and the cutting anastomosis line is carefully checked for integrity and air leakage. if the anastomosis is complete and there is no air leakage, the anastomosis is considered successful.other wise it is considered failed.

SECONDARY OUTCOMES:
operative time | Perioperative/Periprocedural
intra-operative blood loss | Perioperative/Periprocedural
post-operative air leak | Perioperative/Periprocedural
incidence of conversion to open surgery due to stapler-related issues | Perioperative/Periprocedural
complication | Perioperative/Periprocedural

CONTACTS AND LOCATIONS:
Locations (1):
- Jinhua Municipal Central Hospital, Jinhua, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No